CLINICAL TRIAL: NCT06936865
Title: Effectiveness of a Home-Based Multicomponent Exercise Program With Digital Support in Community-Dwelling Older Adults With Falls: A Multicenter Quasiexperimental Trial (GAITCARE Study)
Brief Title: Effectiveness of a Home-Based Multicomponent Exercise Program With Digital Support in Community-Dwelling Older Adults With Falls
Acronym: GAIT2CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish National Research Council (Other Government)
Collaborators: Hospital Universitario Infanta Leonor (Other); Servicio de Salud de Castilla La Mancha, Albacete, Spain (Unknown); Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Antonio R. Jiménez Ruiz, Tenured Scientist, Spanish National Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GAIT2CARE-2023; CEIm approval code 2023-071 (Other: Ethics Committee approval - Hospital Universitario de Albacete (CEIm))
Record Dates: First submitted 2025-04-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Falls; Frailty Syndrome; Gait Disorders; Mobility Limitation; Aging; Sedentary Behaviors
Keywords: Multicomponent Exercise; Digital Health; Home-based Intervention; Older Adults; Physical Performance; VIVIFIL App; Fall Prevention; Remote Monitoring; Geriatric Rehabilitation
MeSH Terms: conditions — Frailty; Mobility Limitation; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This study follows a parallel, non-randomized interventional model. Participants were assigned to one of two arms based on the hospital where they received care, following standard clinical practice. No crossover occurred between groups. Each arm received a multicomponent exercise intervention with similar structure and objectives, delivered either in-person or at home with digital support. The primary comparison focuses on functional outcomes and fall incidence between the two settings.
Masking Description: No masking was implemented. All participants and study personnel were aware of group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Exercise with Digital Support (ViviFil App) (Experimental): Participants in this arm followed a personalized multicomponent exercise program at home using the VIVIFIL mobile application. The program included strength, balance, flexibility, and aerobic exercises adapted to each participant's functional capacity (based on SPPB score). The VIVIFIL App was installed on participants' smartphones or provided devices and included daily video-guided sessions, automatic progression, and a chat function for communication with healthcare professionals who provided remote monitoring.
  Interventions: Behavioral: VIVIFIL App Program
- In-person Supervised Exercise at Geriatric Day Hospital (Active Comparator): Participants in this arm attended supervised multicomponent exercise sessions at the Geriatric Day Hospital, 2-4 times per week for 8 weeks. Each session lasted 45-60 minutes and was delivered by trained professionals. Exercises included strength training, balance exercises, flexibility, and aerobic conditioning. Programs were tailored based on the participant's initial functional assessment.
  Interventions: Behavioral: Hospital-Based Multicomponent Exercise

INTERVENTIONS:
Behavioral: VIVIFIL App Program — A digitally supported multicomponent exercise program delivered through the VIVIFIL mobile application. Participants followed a daily home-based routine including strength, balance, flexibility, and aerobic exercises, adapted to their functional reserve. The app provided video instructions, progression tracking, and a chat for remote communication with healthcare professionals.
  Arms: Home-based Exercise with Digital Support (ViviFil App)
Behavioral: Hospital-Based Multicomponent Exercise — A supervised multicomponent exercise program delivered at a geriatric day hospital by trained professionals. Sessions lasted 45-60 minutes, 2-4 times per week for 8 weeks. Exercises included strength training, balance, flexibility, and aerobic components, adjusted to the participant's functional status.
  Arms: In-person Supervised Exercise at Geriatric Day Hospital

SUMMARY:
This study evaluates the effectiveness of an 8-week multicomponent exercise program conducted at home with digital support through the VIVIFIL mobile application, compared to a traditional in-person hospital-based exercise program, in community-dwelling older adults with a history of falls. The GAIT2CARE study is a multicenter, non-randomized, quasiexperimental clinical trial conducted in three Spanish public hospitals.

Participants aged 70 years or older were assigned to one of two intervention groups depending on the hospital: (1) home-based exercise using the VIVIFIL App with remote monitoring by a healthcare professional, or (2) conventional in-person multicomponent exercise supervised at the hospital. Both interventions included aerobic, strength, balance, and flexibility training.

The study aims to assess improvements in physical performance (SPPB, TUG, gait speed), frailty status, and fall incidence. Baseline and post-intervention assessments were conducted over an 8-week period. The hypothesis is that the home-based digital program is as effective as in-person exercise in improving functional outcomes and preventing falls in older adults.

DETAILED DESCRIPTION:
The GAIT2CARE study is a multicenter, non-randomized, quasiexperimental clinical trial designed to evaluate the effectiveness of a home-based, multicomponent exercise intervention supported by a mobile application (VIVIFIL App) compared to a conventional in-person hospital-based program in community-dwelling older adults with a history of falls.

The study was conducted in three public university hospitals in Spain: Hospital Universitario Infanta Leonor, Hospital Universitario de Getafe, and Hospital Universitario de Albacete. A total of 127 participants aged 70 years or older were recruited from specialized fall clinics between December 2023 and March 2024. Eligibility criteria included a history of falls, ability to walk independently or with one or two canes, and absence of terminal illness. Participants were assigned to either the intervention or control group based on their hospital site, as per standard clinical practice.

The intervention group used the VIVIFIL App, a tool specifically designed for older adults to guide daily exercise at home. The App includes tailored training programs based on functional reserve (measured by SPPB), progressive difficulty levels, and real-time communication with healthcare professionals. Participants who lacked smartphones were provided with one and received training on how to use the App.

The control group attended conventional multicomponent exercise sessions (45-60 minutes, 2-4 times per week) at a geriatric day hospital under professional supervision. Both programs included strength, aerobic, flexibility, and balance training.

Primary outcomes included changes in physical performance (SPPB, Timed Up and Go [TUG], 4-meter gait speed), frailty status, and incidence of falls. Assessments were conducted at baseline and after 8 weeks. The study also included an analysis of factors influencing response to the intervention, such as baseline frailty, cognitive status, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older
* Attending a specialized falls clinic at one of the participating hospitals
* Able to ambulate independently or with the aid of one or two canes
* At least one of the following:

  1. A fall with consequences requiring medical attention in the past year
  2. Two or more falls in the past 12 months
  3. Self-reported gait or balance disturbance
  4. Self-reported fear of falling

Exclusion Criteria:

* Terminal illness with a life expectancy of less than 6 months
* Refusal or inability to provide informed consent

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 127 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Score | Baseline and 8 weeks
  The SPPB is a standardized assessment tool that includes gait speed, chair stand, and balance tests. Scores range from 0 to 12, with higher scores indicating better physical performance. The primary outcome is the change in total SPPB score from baseline to 8 weeks.

SECONDARY OUTCOMES:
Change in 4-Meter Gait Speed | Baseline and 8 weeks
  Gait speed (m/s) is measured over a 4-meter walk. The best of three trials is recorded. Higher speed reflects better functional capacity.

OTHER OUTCOMES:
Change in Timed Up and Go (TUG) Test | Baseline and 8 weeks
  The TUG test assesses functional mobility. Participants are timed as they rise from a chair, walk 3 meters, turn, return, and sit. A lower time indicates better performance.
Change in Frailty Status (Standardised Frailty Criteria) | Baseline and 8 weeks
  Frailty status is assessed using criteria including weight loss, grip strength, exhaustion, slow gait, and low activity. Participants are classified as robust, pre-frail, or frail.
Number of Falls During the Intervention Period | 8 weeks
  Total number of falls reported by participants during the 8-week intervention period. Falls were self-reported and monitored by the research team.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor - HUIL, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) underlying published results will be made available after study completion and publication. The data will be fully anonymized and shared upon reasonable request with qualified researchers for academic and non-commercial purposes. Requests must include a methodologically sound proposal and may require approval by an independent ethics committee. Data access will be provided through a secure platform or encrypted file transfer.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Individual participant data (IPD) and supporting information will be available beginning 6 months after publication of the primary results and will remain accessible for a period of 5 years.
Access Criteria: Qualified researchers affiliated with academic or clinical institutions may request access to anonymized individual participant data (IPD) and supporting documents. Requests must include a scientifically sound research proposal and may require approval by an ethics committee. Data will be shared via secure electronic transfer after signing a data access agreement that ensures confidentiality and appropriate data use.